CLINICAL TRIAL: NCT02718638
Title: Effects of a Program of Strength Physical Activities on the Expression of Nrf2 and Nf-kb Hemodialysis Patients
Brief Title: Effects of Physical Activities on the Expression of Nrf2 and Nf-kb Hemodialysis Patients
Acronym: Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Denise Mafra, Professor, Universidade Federal Fluminense
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeniseMafra2
Record Dates: First submitted 2015-12-01; First posted 2016-03-24 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Chronic Kidney Disease; Hypertension; Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physical exercises group (Other): Physical exercises were performed during HD sessions, at second hour of HD, three times per week for 3 months (36 sessions). The patients remained seated while performing the exercises that were performed in both lower limbs. Ankle-cuffs and elastic bands (Theraband®, Akron-OH, USA) were used for performed the exercises. The physical exercises consisted of four different exercises and they were administered by a physical therapist following the adapted protocol.
  Interventions: Other: physical exercises

INTERVENTIONS:
Other: physical exercises — Physical exercises were performed during HD sessions, at second hour of HD, three times per week for 3 months. The first exercise was knee extension from 90° to 0°. The patient remained in the 0° position for 5 seconds (an isometric contraction) and then returned to the starting position (90º). 2) The second exercise consisted of a triple flexion followed by extension of the lower limbs. The patient flexed the thigh, knee and ankle (elastic band placed at the level of the metacarpals) followed by a double extension of the thigh and knee. 3) In a co-isometric contraction, the patient performed a leg extension against the ankle-cuff resistance (located under the distal third of the leg at the level of the malleolus) for 10 seconds. 4) The patient performed a unilateral hip joint flexion of the lower limb with the knee extended by rising to their functional limit.

SUMMARY:
Oxidative stress and inflammation are cardiovascular risk factors in patients with chronic kidney disease (CKD) undergoing hemodialysis (HD). Nuclear transcription factors play roles in the coordinated expression of genes involved in inflammation, such as nuclear factor Kappa B (NFkB) that increase the cytokines synthesis and Nuclear factor erythroid 2-related factor 2 (Nrf2) that increase the transcription of genes encoding enzymes of phase II detoxifying and antioxidant enzymes. The aim of this study was to evaluate the effects of resistance exercise program on the expression of transcription factors Nrf2 and NF-kB in HD patients.

DETAILED DESCRIPTION:
This study included 44 patients on regular HD program which 25 patients (54.5% women, age 45.7 ± 15.2 years and time on dialysis, 71.2 ± 45.5 months) composed the exercise group and 19 patients (61.5% women, age 42.5 ± 13.5 years and time on dialysis, 70.1 ± 49.9 months) the control group. The exercise program was performed during HD sessions, 3 times a week (36 exercises sessions). Peripheral blood mononuclear cells (PBMC) were isolated and processed for expression of Nrf2, NF-kB and NADPH quinone oxidoreductase 1 (NQO1) by quantitative real-time polymerase chain reaction. Antioxidant enzymes activity (catalase-CAT and glutathione peroxidase-GPx), high-sensitivity C-reactive protein (hs-CRP) and nitric oxide (NO) products were assessed using an enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were age >18 years
* Without any motor skill disorders, arteriovenous fistula for vascular access in the upper limb and patients on maintenance dialysis for at least 6 months.

Exclusion Criteria:

* Patients with autoimmune diseases, cancer, infectious diseases, acquired immunodeficiency syndrome, uncontrolled hypertension, unstable angina, malignant arrhythmias, pregnant, lower limb amputee, history of stroke, neurological or cardiovascular disease (moderate-intensity physical activity is not routinely recommended)
* Taking catabolizing drugs
* Under regular exercise
* Smokers
* Patients who complied with <75 % of the training were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Changes in Nrf2 expression | changes in Nrf2 expression from baseline and 3 months
  analysed by PCR real time
Changes in cytokines plasma levels | changes in cytokines plasma levels from baseline and 3 months
  cytokines plasma levels like interleukin-6, TNF-alpha evaluated by ELISA methods

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639